CLINICAL TRIAL: NCT03462290
Title: Botulinum Toxin Type A Block of the Sphenopalatine Ganglion in Patients With Persistent Idiopathic Facial Pain: a Randomized, Double-blind, Cross- Over, Placebo-controlled Pilot Study
Brief Title: Botox Injections for Patients With Persistent Facial Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 010817-0; 2017-002518-30 (EudraCT Number)
Record Dates: First submitted 2018-02-26; First posted 2018-03-12 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Facial Pain
Keywords: Botulinum Toxins, Type A; Injections; Sphenopalatine Ganglion Block
MeSH Terms: conditions — Facial Pain | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: a randomized, double-blind, cross-over, placebo-controlled pilot study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin (Experimental)
  Interventions: Drug: botulinum toxin type A; Drug: placebo
- placebo (Placebo Comparator)
  Interventions: Drug: botulinum toxin type A; Drug: placebo

INTERVENTIONS:
Drug: botulinum toxin type A — Botulinum toxin type A, powder for solution, 25 international units (IU), injected towards the sphenopalatine ganglion using MultiGuide
  Other Names: botox
Drug: placebo — solution without botulinum toxin A, injected towards the sphenopalatine ganglion using MultiGuide

SUMMARY:
The main objective of this study is to investigate efficacy and safety of injecting botulinum toxin towards the sphenopalatine ganglion using MultiGuide in patients with persistent idiopathic facial pain

ELIGIBILITY:
Inclusion Criteria:

* Persistent Idiopathic Facial Pain fulfilling diagnostic criteria as classified in The International Classification of Headache Disorders, 3rd edition (ICHD-3 beta version) as modified by the authors of this trial. See below.
* Unsatisfactory effect of available treatment methods as evaluated by a neurologist, ENT specialist or maxillofacial surgeon. The patient should have failed treatment with both anticonvulsant as carbamazepine (Tegretol, Carbatrol) and antidepressant as tricyclic antidepressants
* Average Pain intensity ≥4 (0-10) in Numeric Pain Rating Scale (NRS) on the affected side during the 4-week baseline period
* Written informed consent from the patient

Modified diagnostic criteria for PIFP according to The International

Classification of Headache Disorders, 3rd edition (ICHD-3 beta version):

A. Facial and/or oral pain fulfilling criteria B and C.

B. Recurring daily for >2 hr per day for >3 months

C. Pain has both of the following characteristics:

1. Poorly localized and may radiate beyond the trigeminal nerve distribution
2. Dull, aching or nagging quality D. Clinical neurological examination is normal, however patient may denote paresthesia E. A dental cause has been excluded by appropriate investigations; signs of structural pathology or other specific causes of pain are not identified. Minor operation and injury (insignificant trauma e.g. tooth extraction) to the face, maxilla, teeth and gums without a direct causal relationship with the pain regarding both time and site is accepted. F. Not better accounted for by another ICHD-3 diagnosis.

Exclusion Criteria:

* Bilateral symmetrically affected
* Neurological disorders or other related systemic diseases that can explain the pain
* MRI/CT examination confirming intracranial pathology.
* Systemic or local disease or condition that can give a significantly increased risk of complications to the particular procedure
* Not competent to asses informed consent based on neurological assessment
* Psychiatric disorder that prevents the completion of the study
* Pregnancy
* Inappropriate use of contraception
* Breastfeeding
* Abuse or unauthorized use of medication, drugs or alcohol
* Allergy or other hypersensitivity reactions to marcaine, lidocaine, xylocaine, or adrenaline, possibly similar related drugs
* Anatomical factors that prevent or impede the injection
* Known hypersensitivity to botulinum toxin type A or to any of the excipients
* Treatment with drugs that can interact with botulinum toxin type A: aminoglycoside antibiotics, spectinomycin, neuromuscular blockers, both depolarizing (succinylcholine) and non-depolarizing (tubocurarine derivatives), lincosamides, polymyxins, quinidine, magnesium sulfate, anticholinesterases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Changes from baseline to weeks 5-8 in Numeric Pain Rating Scale (NRS) score for persistent idiopathic facial pain (PIFP) | 5-8 weeks
  NRS score for persistent idiopathic facial pain (PIFP) as registered in the pain diary in the active group versus the placebo group. Responders are defined as those with at least 30% reduction in NRS for PIFP in weeks 5- 8 compared to baseline

SECONDARY OUTCOMES:
Percentage of patients with pain intensity rating 1-3 (mild pain) | 8 weeks
Physical functioning assessed by a Multidimensional Pain Inventory or Brief Pain Inventory interference scale | 8 weeks
  the total range of the scale is 10, ranging from 0-10 where 0 is no pain and 10 is worst pain imaginable. No subscale. The higher values the worse outcome.
Physical functioning assessed by Norwegian Pain association - minimal questionnaire (NOSF-MISS) | 8 weeks
Quality of life according to Questionnaire for quality of life, Patient Global Impression of Change (PGIC) | 8 weeks
Number of days without persistent idiopathic facial pain | 8 weeks
number of doses of analgesics per 4 weeks | 8 weeks
Sick leave due to persistent idiopathic facial pain | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, PhD prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Neuroscience, Faculty of Medicine and Health Science, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jamtoy KA, Thorstensen WM, Stovner LJ, Rosen A, Maarbjerg S, Bratbak D, Simpson MR, Tronvik E. Onabotulinum toxin A block of the sphenopalatine ganglion in patients with persistent idiopathic facial pain: a randomized, triple-blind, placebo-controlled, exploratory, cross-over study. Cephalalgia. 2023 Jul;43(7):3331024231187132. doi: 10.1177/03331024231187132. PMID 37435807